CLINICAL TRIAL: NCT00226616
Title: Clinical Trial of Zinc Supplementation in Cholera Patients
Brief Title: Zinc Supplementation in Cholera Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Thrasher Research Fund (Other); World Bank (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 99-022
Record Dates: First submitted 2005-09-25; First posted 2005-09-27 (Estimated); Last update posted 2005-10-20 (Estimated); Status verified 2005-09

CONDITIONS: Cholera
Keywords: Zinc; cholera; children; Bangladesh
MeSH Terms: conditions — Cholera | interventions — Zinc

INTERVENTIONS:
Drug: Zinc

SUMMARY:
Cholera is one of the leading causes of morbidity and mortality among children and adult in developing countries. We will evaluate the effect of supplementation of zinc on reduction of duration and severity of cholera. Since cholera is primarily a disease of older children and adults, we intend to study the effects of zinc supplementation among children of 3 to 14 years of age, whose initial stool weight will be >4ml/kg/hour in 1st 6 hours and dark field examination is positive. 90 subjects in each group hospitalized with cholera with diarrhea for less than 24 hours will be selected. After inclusion in the study, informed consent will be obtained from guardian explaining the full procedure in the hospital. The subjects will be randomized to receive either zinc or placebo until diarrhea resolves. History of illness and baseline information will be collected in the hospital through interview, which may take duration of 10 minutes.After 6 hours of initial rehydration, fluid balance study will be carried out on all subjects until diarrhea resolves. 1 ml (1/4 teaspoonful) of blood sample will be taken to assess serum zinc level on admission after initial hydration and will be repeated on the day of recovery. This procedure carries a small risk of infection if not done under sanitary conditions; however, we will maintain proper sanitation, so there is no risk in the procedures. There is no potential risk in this study.20mg elemental Zinc will be given daily in 2 divided doses till cholera resolves. Both groups will receive syrup or tablet Erythromycin 50mg/kg/24 in 4 divided doses for 3 days. Oral rehydration solution/intravenous acetate fluid will be used for rehydration. Daily body weight will be taken and stool will be sent for C/S until the day of recovery or 5 days. Zinc loss in stool will be seen in 20% of random stool samples. Information obtained from history and the laboratory investigations of subject will be kept strictly confidential and no one other than the investigators of this study and the Ethics Committee of this Centre will/ has access to the information. The study will benefit the patients as study physician will do close observation, examination and will take care frequently, as research staff will monitor systematic progress and take necessary action. Study micronutrient (zinc) is shown to have benefit in children in acute diarrhea. If the results of the study is positive, it will benefit the patients in their treatment during this study and thereafter. The data will be analyzed for clinical effects of zinc on diarrhea.The study will help to improve the treatment strategy of cholera in children. The study will use hospital records, which will be returned after completion of the study. Stool, urine and 1 ml (1/4 teaspoonful) of venous blood will be taken to assess serum zinc level.

DETAILED DESCRIPTION:
Study design:

A double blind randomized clinical trial using zinc and placebo.

Randomization:

Patients will be randomized to one of two groups, A or B. Block randomization will be done using block length of 6. Group A will receive Zinc+ Erythromycin and Group B: will receive Placebo+Erythromycin

Dose of Erythromycin

Syrup/tab Erythromycin 50mg/kg/24 hours in 4 divided doses for 3 days.

Dose of zinc:

Zinc acetate will be given at 10mg twice daily (10mgx2=20mg elemental zinc) until cholera resolves (the time of passage of last unformed stool or first formed stool followed by 24 hours without any diarrheal stool).

Composition of the syrup:

For both groups, the bulk of the base syrup will be consist of the same chemicals; in addition to this, group A will have the treatment substance (i.e. elemental zinc 20 mg/day)

Syrup A: Quantity per 5 ml

Zinc Acetate 10 mg elemental zinc

Syrup B: Base substance

Base Substance:

Ascorbic acid 30 mg Glycerin USP 1.2 ml Propylene glycol USP 0.75 ml Sorbitol 70% BP 2.0 ml Methyl Paraben USFN 3.5 mg Polysorate-80 50 mg (Tween -80) BPC Lemon oil PH grade 0.0125 ml Caramel Brown colour 1 mg Purified water 0.75 ml

Clinical procedure in the hospital:

Patients who meet the selection criteria will be observed for initial six hours, while their urine and stool specimen will be collected separately. Patient whose initial stool-output >4ml/kg/hour during this period and dark field examination of stool is positive will be enrolled in the study. Patients will be kept in study ward. After complete hydration, patients will be randomised in blocks of 6 to one of two groups A and B. Group A will receive syrup zinc and group B will receive placebo till cholera resolves. Both the groups will receive the identical bottles containing syrup with same flavor and only single unique serial number will be written on the bottles. The number will indicate an exact subject of study. Both the groups will receive Syrup/Tab Erythromycin. 1ml blood will be collected for serum zinc on admission after complete dehydration and this test will be repeated at the time of discharge. Stool culture and sensitivity (C/S) will be sent daily until the day of recovery or 5 days. Balance will be performed on all the patients till cholera resolves. If any complication develops after enrollment, study will be discontinued and patient will be treated accordingly.

Assessment of dehydration:

To reduce observational variation, especially regarding the assessment of dehydration, a standardized form is developed for the assessment of dehydration.

CONDITION* (1=normal, 2=irritable/lessactive, 3=lethargic/comatose) MUCOSA (1=normal, 2=dry)

EYES (1=normal, 2=sunken) THIRST* (1=normal, 2=thirsty, 3=unable to drink) SKIN TURGOR* (1=normal, 2=reduced) PULSE* (1=normal, 3=feeble/absent)

DEHYDRATION STATUS:

1. no sign of dehydration
2. some dehydration (two signs coded 2 with at least one key sign*)
3. severe dehydration (some dehydration, plus one key sign* coded 3)

(* This method was recently validated by a group of international experts in oral rehydration therapy who were invited to ICDDR, B and is currently being used in a large WHO sponsored multi-centre trial for the evaluation of low osmolarity ORS. The investigators have been trained in this method).

Rehydration phase:

All the patients recruited in this study, will have either, some dehydration or severe dehydration. Therefore, before being randomized into study, during initial 6 hours all the patients will be rehydrated either by ORS or intravenous fluid. Patients with signs of some dehydration will be rehydrated by ORS and patients with severe dehydration will be rehydrated intravenously as described below. The following IV fluids will be used:

Sodium Potassium Chloride Acetate Dhaka Solution (mmol/L) (mmol/L) (mmol/L) (mmol/L) 133 13 98 48 Rate of administration will be 100 ml/kg over 4 hours, plus volume-for-volume replacement for ongoing losses hourly.

If, at the end of four hours:

1. The patient is fully rehydrated, he/she will be randomized to one of the treatment groups;
2. Some dehydration persist, IV infusion will continue at the rate of 50 ml /kg over 2 hours, plus replacement volume for volume of ongoing losses;
3. Severe dehydration persists, IV infusion will continue for an additional 2 hours at the rate of 100 ml/kg, plus replacement of ongoing losses. This is very unusual, however, occurring only in very few patients who pass large watery stools frequently.

If at the end of six hours, the patient is fully rehydrated patient will be randomized to one of the treatment group. If signs of dehydration persist after 6 hours, the patient will be excluded from study. All intake and output during this initial rehydration phase will be recorded.

Maintenance phase:

After completion of rehydration, subjects will be randomized to one of the two groups Group A and Group B. Group A will be given zinc acetate and group B will be given placebo. The supplementation of zinc or placebo will be continued till diarrhea resolves. Ongoing stool losses will be replaced with equal volume of Rice-ORS.

Dietary management:

Standardize hospital diet will be given to all patients which includes milk suji, rice, vegetable, daal, bread banana and chicken or fish.

Intake and output measurement:

All oral and intravenous fluid will be measured and recorded until cholera resolves. Stool weight will be measured separately from urine every 8 hours until cholera resolves. Urine will be separated and measured 8 hourly, weight of vomitus will also be taken 8 hourly. Daily clinical examination will be done by the investigators and study physician with observation on stool consistency and character.

Clinical recovery:

Clinical recovery will be defined as the time of passage of last unformed stool or first formed stool followed by 24 hours without any diarrheal stool.

Sample size calculation:

We assume that zinc will reduce 20% of mean duration of illness compared to erythromycin group18 at 90% power and 5% level of confidence. Therefore the sample size will be:

n=2 (SD)2 aß/(D)2 n=2 (5)2 10.5/(2.6)2 n=77.66=78 per treatment group So the total number of samples will be 78 x 2 =156. Considering 15% drop out the total number of samples will be 156+24=180

Assessment of weight gain:

Weight will be taken on admission and daily until cholera resolves.

Laboratory tests:

1. Microscopic examination

   1. Dark field examination will be done on stool samples on admission.
2. Microbiological assays:

   1 Daily stool C/S will be done till cholera resolves or 5 days.
3. Micronutrient assay:

   1. Serum zinc level will be obtained on day 1 and on the day of recovery
   2. Randomly zinc loss in cholera will be seen in 20% samples.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 3-14 years hospitalized at ICDDR, B presenting with cholera within 24 hours of onset.
* Stool output more than 4ml/kg/hour within the first 6 hours of observation period.
* Positive dark field examination

Exclusion Criteria:

* Unable to rehydrate within 6 hours
* Negative dark field examination
* Systemic illness requiring immediate administration of antibiotics.
* Received antibiotics in the 24 hours prior to hospitalization
* Patients presenting with bloody mucoid diarrhea
* Unconscious or medical emergencies

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2000-11; Study Completion 2002-07

PRIMARY OUTCOMES:
Reduction in duration of diarrhoea
Reeudction in total stool volume

SECONDARY OUTCOMES:
Serum Zinc status

CONTACTS AND LOCATIONS:
Overall Officials: Swapan K Roy, MBBS,MSc,Phd, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (2):
- Bangladesh (2):
  - ICDDR,B, Dhaka hospital, Dhaka
  - S.k.Roy, Dhaka

REFERENCES:
- [Derived] Roy SK, Hossain MJ, Khatun W, Chakraborty B, Chowdhury S, Begum A, Mah-e-Muneer S, Shafique S, Khanam M, Chowdhury R. Zinc supplementation in children with cholera in Bangladesh: randomised controlled trial. BMJ. 2008 Feb 2;336(7638):266-8. doi: 10.1136/bmj.39416.646250.AE. Epub 2008 Jan 8. PMID 18184631